CLINICAL TRIAL: NCT03278860
Title: The Effects of Intranasal Oxytocin on Social Touch: an fMRI-based Study
Brief Title: The Effects of Oxytocin on Social Touch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-39
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Oxytocin; social touch

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind within-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin then placebo (Experimental): Participants first received oxytocin (24 IU). After a washout period of 2 weeks, they then received placebo (24 IU).
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo
- Placebo then oxytocin (Experimental): Participants first received placebo (24 IU). After a washout period of 2 weeks, they then received oxytocin (24 IU).
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo

INTERVENTIONS:
Drug: intranasal oxytocin — 24 IU of oxytocin nasal spray will be applied to each subject.
  Arms: Oxytocin then placebo
Drug: intranasal placebo — an identical amount of placebo nasal spray will be applied to each subject.
  Arms: Oxytocin then placebo
Drug: intranasal oxytocin — 24 IU of oxytocin nasal spray will be applied to each subject.
  Arms: Placebo then oxytocin
Drug: intranasal placebo — an identical amount of placebo nasal spray will be applied to each subject.
  Arms: Placebo then oxytocin

SUMMARY:
The main aim of the study is to investigate whether intranasal oxytocin (24IU) can enhance hedonic experience and associated brain-reward reward responses to social touch.

DETAILED DESCRIPTION:
A double-blind, within-subject, placebo controlled design is employed in this study. In total 50 healthy male subjects will be recruited and they will come twice, once with the administration of oxytocin nasal spray and the other placebo (interval time is more than 2 weeks). 45 minutes after treatment subjects will be applied two different types of pleasant touch: social touch from a masseur (professional therapist) and non-social touch from a massage device. After each condition the subjects will be asked to rate pleasantness, likability, and arousal. Simultaneously functional brain activity will be acquired via fMRI. Blood samples will be taken before and after the intervention to assess oxytocin levels. All subjects were asked to complete a range of questionnaires measuring trait personality and mood: Beck Depression Inventory (BDI), Cheek and Buss Shyness Scale (CBSS),Autism Spectrum Quotient (ASQ), Empathy Quotient (EQ), NEO Five Factor Inventory (NEO-FFI), Liebowitz Social Anxiety Scale (LSAS),Behavioral Inhibition System and Behavioral Activation System Scale (BISBAS),Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ),State-Trait Anxiety Inventory (STAI), Social Touch Questionnaire (STQ), Sensory over Responsivity Scale (SOR) and Under Responsivity Scale (URS) one day before the first scanning. On the first and second scanning day, the subjects were asked to complete Positive and Negative Affect Schedule (PANAS) before and after treatment administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury
* Medical or mental illness

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Neural indices: fMRI-based measures of interoceptive and reward processing | 45-90 minutes after treatment administration
  fMRI-based measures of social and non-social touch-related brain activity

SECONDARY OUTCOMES:
Behavioral index: pleasantness experience | 45-90 minutes after treatment administration
  Ratings for pleasantness during the application of social and non-social touch
Behavioral index: likability experience | 45-90 minutes after treatment administration
  Ratings for likability during the application of social and non-social touch
Behavioral index: arousal experience | 45-90 minutes after treatment administration
  Ratings for arousal during the application of social and non-social touch

CONTACTS AND LOCATIONS:
Overall Officials: Qin Li, MA, Study Chair — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China

REFERENCES:
- [Derived] Chen Y, Li Q, Zhang Q, Kou J, Zhang Y, Cui H, Wernicke J, Montag C, Becker B, Kendrick KM, Yao S. The Effects of Intranasal Oxytocin on Neural and Behavioral Responses to Social Touch in the Form of Massage. Front Neurosci. 2020 Dec 4;14:589878. doi: 10.3389/fnins.2020.589878. eCollection 2020. PMID 33343285